CLINICAL TRIAL: NCT01787513
Title: A Randomised Controlled Trial Comparing Internet Based Cognitive Behavioural Therapy for Major Depressive Disorder Plus a Cognitive Bias Modification Intervention (OxIGen)on Symptoms of Depression and Negative Interpretation Bias.
Brief Title: Cognitive Bias Modification (CBM) Via Imagery and Internet Cognitive Behavioural Therapy (iCBT) for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Alishia Williams, Principal Investigator, St Vincent's Hospital, Sydney
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/237
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBM Version A + iCBT (Experimental): CBM Version A is an Internet-based intervention taking place over 1 week followed by iCBT, an Internet-based treatment for depression taking place over 10 weeks.
  Interventions: Other: CBM; Other: iCBT
- CBM Version B (Control) + iCBT (Placebo Comparator): CBM Version B (Control) is an Internet-based intervention taking place over 1 week (identical to CBM Version A without the putative active components) followed by iCBT, an Internet-based treatment for depression taking place over 10 weeks.
  Interventions: Other: CBM; Other: iCBT

INTERVENTIONS:
Other: CBM — CBM is an Internet-based intervention comprised of delivery of auditory scenarios taking place over 1 week.
Other: iCBT — iCBT is a validated online CBT treatment program for depression delivered in 6 lessons over 10 weeks.

SUMMARY:
A randomised controlled trial comparing Internet based cognitive behavioural therapy for major depressive disorder plus a cognitive bias modification intervention (OxIGen) version A vs. Internet based cognitive behavioural therapy for major depressive disorder plus a cognitive bias modification intervention (OxIGen) version B on symptoms of depression and negative interpretation bias.

DETAILED DESCRIPTION:
Cognitive accounts of depression and anxiety emphasize the importance of cognitive biases in the maintenance of disorders. One specific bias is the interpretation of ambiguous information. A negative interpretation bias is defined as a systematic tendency to interpret potentially ambiguous information in a negative rather than benign way and this bias has been associated with symptoms of depression. Research has led to the recent development of computerized cognitive bias modification (CBM) techniques to augment such biases and it has been suggested that CBM techniques may be useful as an adjunct to current treatments to enhance maintenance of treatment gains and minimize relapse rates. The fact that CBM procedures lend themselves to being delivered remotely, are cost-effective, and can be self-paced in ways that suit the patient make them an ideal candidate for inclusion in the Internet-based cognitive behavioural therapy (iCBT) programs currently offered through St. Vincent's Hospital and the University of New South Wales. Therefore, the primary aim of the current trial is to evaluate the acceptability and effectiveness of adding CBM procedures to the existing iCBT modules offered through St. Vincent's Hospital and the University of New South Wales. It is expected that iCBT + CBM (active version) will result in superior treatment outcomes as indexed by a standardized clinical battery compared to iCBT + CBM (control version).

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of the American Psychiatric Association - 4th edition (DSM-IV) criteria for Major Depressive Disorder
* Internet and printer access
* Australian resident
* Fluent in written and spoken English

Exclusion Criteria:

* Current substance abuse/dependence
* Psychotic mental illness (Bipolar or Schizophrenia)
* Change in medication or psychological treatment during last 1 month or intended change during study duration
* Use of Benzodiazepines
* Severe depression (PHQ9> 23)
* Suicidal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9)scores | Administered at baseline (T1), post-CBM intervention (T2, 1 week after baseline), post iCBT intervention (8-10 weeks after baseline), and at 3 month follow-up (T4).
Change in Beck Depression Inventory - second edition (BDI-II)scores | Administered at baseline (T1), post-CBM intervention (T2, 1 week after baseline), post iCBT intervention (8-10 weeks after baseline), and at 3 month follow-up (T4).
Change in Ambiguous Sentence Task (AST)scores | Administered at baseline (T1), post-CBM intervention (T2, 1 week after baseline).
Change in diagnostic status (MINI5 depression module) | Administered at baseline (T1), post iCBT intervention (8-10 weeks after baseline), and at 3 month follow-up (T4).

SECONDARY OUTCOMES:
Change in Kessler-10 (K10)scores | Administered at baseline (T1), post-CBM intervention (T2, 1 week after baseline), post iCBT intervention (8-10 weeks after baseline), and at 3 month follow-up (T4).
Change in WHO Disability Assessment Scale (WHO-DAS)scores | Administered at baseline (T1, post iCBT intervention (8-10 weeks after baseline), and at 3 month follow-up (T4).
Change in State Trait Anxiety Inventory (STAI)scores | Administered at baseline (T1), post iCBT intervention (8-10 weeks after baseline), and at 3 month follow-up (T4).
Change in Repetitive Thinking Questionnaire (RTQ)scores | Administered at baseline (T1), post-CBM intervention (T2, 1 week after baseline), post iCBT intervention (8-10 weeks after baseline), and at 3 month follow-up (T4).
Change in Clinical Perfectionism Scale (PCS)scores | Administered at baseline (T1), post iCBT intervention (8-10 weeks after baseline), and at 3 month follow-up (T4).

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Andrews, MD, Principal Investigator — UNSW; ST. Vincent's Hospital; Alishia Williams, PhD, Principal Investigator — UNSW; ST Vincent's Hospital
Locations (1):
- St. Vincent's Hospital, Darlinghurst, New South Wales, Australia

REFERENCES:
- [Derived] Williams AD, Blackwell SE, Holmes EA, Andrews G. Positive imagery cognitive bias modification (CBM) and internet-based cognitive behavioural therapy (iCBT) versus control CBM and iCBT for depression: study protocol for a parallel-group randomised controlled trial. BMJ Open. 2013 Oct 29;3(10):e004049. doi: 10.1136/bmjopen-2013-004049. PMID 24171941